CLINICAL TRIAL: NCT02881385
Title: Effects on Respiratory Patterns and Patient-ventilator Synchrony in Different Ventilator Using Pressure Support Ventilation
Brief Title: Effects on Respiratory Patterns and Patient-ventilator Synchrony Using Pressure Support Ventilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, physician, Southeast University, China
Other Study IDs: zhongdayiyuanICU
Record Dates: First submitted 2016-07-30; First posted 2016-08-29 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Acute Respiratory Distress Syndrome; COPD; Post Operative
Keywords: Synchrony; Pressure Support Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- E5 Esense 10%: PSV mode using E5 ventilator with Esense 10%
- E5 Esense 30%: PSV mode using E5 ventilator with Esense 30%
- E5 Esense 50%: PSV mode using E5 ventilator with Esense 50%
- Servo-I Esense 10%: PSV mode using Servo-I ventilator with Esense 10%
- Servo-I Esense 30%: PSV mode using Servo-I ventilator with Esense 30%
- Servo-I Esense 50%: PSV mode using Servo-I ventilator with Esense 50%
- E5 Esense autocycle: PSV mode using E5 ventilator with Esense Auto cycle

SUMMARY:
Pressure Support Ventilation use Expiratory triggering sensitivity(Esense) to transfer inspiration to expiration,the value of Esense is fixed.That may lead to asynchrony between humans and ventilators,making people uncomfortable and prolonging weaning time.Some ventilators have auto cycle function Based on curves of pressure on respiratory patterns,it will make the transforming more synchrony with humans.Our prospective observational study will prove the superiority of the auto cycle function.

DETAILED DESCRIPTION:
From August 31st 2016 to August 31st 2017, all ARDS 、COPD and postoperative patients admitted to the ICUs will be enrolled. The demographic characteristics, diagnosis, formerly medical history, Ventilator indications, Ventilator data, other respiratory treatments, weaning outcome and 28 day mortality will be recorded

ELIGIBILITY:
Inclusion Criteria:

ARDS,COPD and Postoperative patient

Exclusion Criteria:

variety of reasons can not be placed next to the bed by the nasal EAdi catheter

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanical ventilation adult people using PSV mode in ICU
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
patient-ventilator synchrony using PSV mode between different ventilator for 180mins | 180mins after the patients involved

SECONDARY OUTCOMES:
Patient Respiratory Patterns during Pressure Support Ventilation for 180mins | 180mins
Patient gas exchange during Pressure Support Ventilation for 180mins | 180mins
Effects on Respiratory Patterns in different Expiratory triggering sensitivity for 180mins | 180mins
work of triggering and respiratory in different Expiratory triggering sensitivity for 180mins | 180mins

IPD SHARING:
Plan to Share IPD: Undecided